CLINICAL TRIAL: NCT03605537
Title: Use of Mometasone Eluting Stent in Choanal Atresia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to lack of funding.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-1813
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Choanal Atresia
MeSH Terms: conditions — Choanal Atresia | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stent (Experimental): Subjects will undergo repair of the choanal atresia in the operating room with a drug eluting stent placed at the end of the surgical procedure. They will return to the operating room in 3-5 weeks for repeat nasal endoscopy with possible balloon dilation, which is standard of care within our institution. At this time in the operating room the intervention arm will have the stent removed. Following removal of the stent, photodocumentation of the posterior nasal cavity and nasopharynx will take place to assess the size (standard of care).
  Subjects will then follow up and undergo a bedside or outpatient nasal endoscopy and nasopharyngoscopy (standard of care) at the following approximate intervals 1 month, 6 months, 12 months (these are not exact time periods as clinic scheduling can sometimes be 2-3 months on either side of these time stamps).
  Interventions: Drug: Drug-eluting Stent Mometasone
- No Stent (No Intervention): Subjects will undergo repair of the choanal atresia in the operating room with no stent placed at the end of the surgical procedure. They will return to the operating room in 3-5 weeks for repeat nasal endoscopy with possible balloon dilation, which is standard of care within our institution. Photodocumentation of the posterior nasal cavity and nasopharynx will take place to assess the size (standard of care).
  Subjects will then follow up and undergo a bedside or outpatient nasal endoscopy and nasopharyngoscopy (standard of care) at the following approximate intervals 1 month, 6 months, 12 months (these are not exact time periods as clinic scheduling can sometimes be 2-3 months on either side of these time stamps).

INTERVENTIONS:
Drug: Drug-eluting Stent Mometasone — The subject will have a mometasone drug-eluting stent placed during their choanal atresia repair procedure instead of no stent being placed.
  Other Names: Mometasone
  Arms: Stent

SUMMARY:
This study is to find out how well drug-eluting stents work as part of treatment for choanal atresia repair. Participants will be receiving surgical choanal atresia repair; half will get a drug-eluting stent placed, the other half will not.

DETAILED DESCRIPTION:
Objective: To determine the utility of mometasone eluting stents in the treatment of choanal atresia.

Setting: Cincinnati Children's Hospital Medical Center (CCHMC), Division of Pediatric Otolaryngology, Head and Neck Surgery

Study Design: Randomized, single blind control trial

Methods: This study will be a randomized, prospective single-blinded control trial. Inclusion criteria will include all subjects less than 11 years of age who are diagnosed with either unilateral or bilateral choanal atresia. Following enrollment, the patients will be randomized to either a control arm (no stent) versus an intervention arm (placement of drug eluting stent). Subjects will then undergo surgical repair of the choanal atresia with either no stent or a drug eluting stent placed. Multiple postoperative nasal endoscopies will be performed to assess size which will be reviewed and graded by two independent reviewers.

Analysis: Descriptive statistical analysis and multivariate analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are under 11 years old and have a diagnosis of choanal atresia will be included in this study.

Exclusion Criteria:

* Those subjects who are 11 years of age or greater or who do not have choanal atresia will be excluded.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Posterior Nasal Cavity | 12 Months
  Once photodocumentation from followup visits is collected, the images will be collected by a member of the team and given to two independent expert blinded reviewers for assessment of the size of the posterior nasal cavity. The picture will be obtained from the same anatomical position for each scope (the posterior portion of the inferior turbinate) and compared to the picture immediately after surgery of the posterior nasal cavity to assess any changes in size. Reviewers will assess the size of the posterior nasal cavity in each subsequent scope and categorize subjects based on the following sizes (0-50%, 51-75%, 76-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Hart, MD, Principal Investigator — CCHMC
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be retained in an identifiable state in a password protected database for potential unspecified research. If this data were to be used in the future, a new IRB would be submitted.

REFERENCES:
- [Background] Deutsch E, Kaufman M, Eilon A. Transnasal endoscopic management of choanal atresia. Int J Pediatr Otorhinolaryngol. 1997 May 4;40(1):19-26. doi: 10.1016/s0165-5876(96)01486-3. PMID 9184974
- [Background] Strychowsky JE, Kawai K, Moritz E, Rahbar R, Adil EA. To stent or not to stent? A meta-analysis of endonasal congenital bilateral choanal atresia repair. Laryngoscope. 2016 Jan;126(1):218-27. doi: 10.1002/lary.25393. Epub 2015 May 25. PMID 26014684
- [Background] Murr AH, Smith TL, Hwang PH, Bhattacharyya N, Lanier BJ, Stambaugh JW, Mugglin AS. Safety and efficacy of a novel bioabsorbable, steroid-eluting sinus stent. Int Forum Allergy Rhinol. 2011 Jan-Feb;1(1):23-32. doi: 10.1002/alr.20020. Epub 2011 Feb 8. PMID 22287304
- [Background] Bangiyev JN, Govil N, Sheyn A, Haupert M, Thottam PJ. Novel Application of Steroid Eluting Stents in Choanal Atresia Repair: A Case Series. Ann Otol Rhinol Laryngol. 2017 Jan;126(1):79-82. doi: 10.1177/0003489416671533. Epub 2016 Oct 7. PMID 27913724
- [Background] Wilcox LJ, Smith MM, de Alarcon A, Epperson M, Born H, Hart CK. Use of Steroid-Eluting Stents after Endoscopic Repair of Choanal Atresia: A Case Series with Review. Ann Otol Rhinol Laryngol. 2020 Oct;129(10):1003-1010. doi: 10.1177/0003489420928374. Epub 2020 May 29. PMID 32468891
- [Background] Schenkel EJ, Skoner DP, Bronsky EA, Miller SD, Pearlman DS, Rooklin A, Rosen JP, Ruff ME, Vandewalker ML, Wanderer A, Damaraju CV, Nolop KB, Mesarina-Wicki B. Absence of growth retardation in children with perennial allergic rhinitis after one year of treatment with mometasone furoate aqueous nasal spray. Pediatrics. 2000 Feb;105(2):E22. doi: 10.1542/peds.105.2.e22. PMID 10654982